CLINICAL TRIAL: NCT01346865
Title: A Randomized, Placebo Controlled, Double-blind, Phase 4 Study to Evaluate Efficacy and Safety of Triple Anti-platelet Therapy Compared With Dual Antiplatelet Therapy in Patients Treated With Drug Eluting Stent for Coronary Artery Disease
Brief Title: Drug-Eluting Stenting Followed by Cilostazol tREAtment Reduces SErious Adverse Cardiac Events (DECREASE-PCI)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: Seung-Jung Park (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, M.D., Ph.D.,Professor of Medicine Asan Medical Center, University of Ulsan, College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVRF2010-10
Record Dates: First submitted 2011-04-22; First posted 2011-05-03 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: triple anti-platelet therapy; dual antiplatelet therapy; DES; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cilostazol (Experimental): cilostazol 100mg
  Interventions: Drug: Cilostazol
- dual therapy group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100mg bid
  Other Names: Pletaal
  Arms: cilostazol
Drug: Placebo — Placebo 1tablet bid
  Arms: dual therapy group

SUMMARY:
The DECREASE-PCI trial is a prospective, randomized, placebo controlled, double-blind, phase 4 study to evaluate efficacy and safety of triple anti-platelet therapy compared with dual antiplatelet therapy in patients treated with DES for Coronary Artery Disease.

The primary objective of this study is to compare the safety and efficacy of triple antiplatelet therapy versus dual (standard) antiplatelet therapy in patients treated with drug-eluting stent (DES) implantation for the treatment of coronary artery disease.

DETAILED DESCRIPTION:
Use of drug-eluting stent (DES) has reduced the incidence of restenosis rate and the need for repeat revascularization compared to using bare metal stents (BMS). Therefore, DES implantation has been default strategy in the treatment of coronary artery disease. However, despite use of DES, the restenosis, subsequent repeat revascularization, and associated cardiac events (stent thrombosis, myocardial infarction) remain significant clinical problem in routine practice, especially complex lesion subsets.

2110 patients who received successful dug eluting stent implantation will be enrolled at 21 centers in Korea. Patients meeting inclusion criteria without any exclusion criteria and agree to participate in this trial will be randomized 1:1 to a) triple therapy (Aspirin+Clopidogrel +Cilostazol) or b) dual therapy group (Aspirin+ Clopidogrel +Placebo). All patients will be blindly assigned to cilostazol 100mg (1tablet bid) or matching placebo (1tablet bid) as 1:1 ratio and are prescribed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical

1. Patients with angina and documented ischemia or patients with documented silent ischemia
2. Patients who are eligible and has been successfully applied for DES implantation
3. Age >18 years
4. Signed written informed consent form prior to study entry

2. Angiographic

1. De novo lesion or restenotic lesions
2. Percent diameter stenosis ≥50%
3. Reference vessel size 2.5 mm by visual estimation

Exclusion Criteria:

1. History of bleeding diathesis or coagulopathy (e.g. current use of NSAIDs, Upper GI bleeding during the recent 6 months)
2. Pregnancy or lactation (women who have child-bearing potential)
3. Known hypersensitivity or contra-indication to contrast agent, heparin, eluted-drug of stent
4. Limited life-expectancy (less than 1 year) due to combined serious disease
5. Characteristics of lesion 1)Left main disease 2)Graft vessels
6. Hematological disease (Neutropenia <3000/mm3, Thrombocytopenia <100,000/mm3)
7. Hepatic dysfunction, liver enzyme (ALT and AST) elevation 3 times normal
8. Renal dysfunction, creatinine 2.0mg/dL
9. Contraindication to aspirin, clopidogrel or cilostazol
10. Stroke (ischemic or hemorrhagic) or transient ischemic attack (TIA) within 6 months.
11. Planned major surgery within the next 6 months with the need to discontinue antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2011-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Ischemic Events (MACCE) | At 1-year time point after PCI
  composite of any death, myocardial infarction, ischemic stroke, target vessel revascularization

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | At 1-year time point and yearly up to 3 years after PCI
  1. Composite of major cardiac adverse events (MACE) including death, Q-MI, Non Q- MI, and target lesion or vessel revascularization
  2. Target vessel revascularization
  3. Target lesion revascularization
  4. Stent thrombosis (definite/probable)
  5. Ischemic stroke
  6. Myocardial infarction
  7. Adverse Events during study periods

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center University of Ulsan College of Medicine
Locations (12):
- South Korea (12):
  - Sejong General Hospital, Bucheon-si
  - Soonchunhyang Univ. Bucheon Hospital, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Pusan National University Yangsan Hospital, Pusan
  - Department of Medicine, Asan Medical Center University of Ulsan College of Medicine, Seoul
  - Gangnam Severance Hospital, Seoul
  - SMA-SNU Boramae Medical Center, Seoul
  - St.carollo Hospital, Suncheon